CLINICAL TRIAL: NCT04480827
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Aramchol in Subjects With Hepatic Impairment
Brief Title: Open-Label Study to Evaluate the Safety, Tolerability, and PK of Aramchol in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Research and Development, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Galmed Pharmaceuticals Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aramchol-019
Record Dates: First submitted 2020-06-02; First posted 2020-07-21 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2022-09

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetics
MeSH Terms: interventions — Salts; Meglumine; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: Mild Hepatic Impairment (Cohort A) (Experimental): 8 mild hepatic impaired subjects
  Interventions: Drug: Aramchol free acid tablet 600mg, single dose
- Part 1: Moderate Hepatic Impairment (Cohort B) (Experimental): 8 moderate hepatic impaired subjects
  Interventions: Drug: Aramchol free acid tablet 600mg, single dose
- Part 1: Severe Hepatic Impairment (Cohort C) (Experimental): 8 severe hepatic impaired subjects
  Interventions: Drug: Aramchol free acid tablet 600mg, single dose
- Part 1: Healthy Volunteers (Cohort D) (Experimental): 15 matched healthy volunteers
  Interventions: Drug: Aramchol free acid tablet 600mg, single dose
- Part 2: Mild Hepatic Impairment Cohort (Experimental): 4 mild hepatic impaired subjects
  Interventions: Drug: Aramchol free acid tablet 300mg, bid
- Part 2: Moderate Hepatic Impairment Cohort (Experimental): 7 moderate hepatic impaired subjects
  Interventions: Drug: Aramchol free acid tablet 300mg, bid
- Part 2: Healthy Volunteers Cohort (Experimental): 7 matched healthy volunteers
  Interventions: Drug: Aramchol free acid tablet 300mg, bid

INTERVENTIONS:
Drug: Aramchol free acid tablet 600mg, single dose — Aramchol free acid tablet 600mg, single dose
  Other Names: Cholan-24-oic acid 7,12-dihydroxy3-[(1- oxoeicosyl)amino]-(3β,5β,7α,12α) salt with N-methyl-(D)-glucamine
  Arms: Part 1: Healthy Volunteers (Cohort D); Part 1: Mild Hepatic Impairment (Cohort A); Part 1: Moderate Hepatic Impairment (Cohort B); Part 1: Severe Hepatic Impairment (Cohort C)
Drug: Aramchol free acid tablet 300mg, bid — Aramchol acid tablet 300mg, bid for 12 days
  Other Names: Cholan-24-oic acid 7,12-dihydroxy3-[(1- oxoeicosyl)amino]-(3β,5β,7α,12α) salt with N-methyl-(D)-glucamine
  Arms: Part 2: Healthy Volunteers Cohort; Part 2: Mild Hepatic Impairment Cohort; Part 2: Moderate Hepatic Impairment Cohort

SUMMARY:
Phase 1, multicenter, open-label, 2-part, single- and multiple-dose study designed to assess the effect of hepatic insufficiency on the PK of aramchol

DETAILED DESCRIPTION:
Each of the 2 parts of the study consisted of a screening period, a check in day, a treatment period, and an end of study (EOS) visit.

In Part 1 (single-dose): 39 subjects were enrolled: 8 subjects each in the mild (Cohort A), moderate (Cohort B), and severe (Cohort C) hepatic impairment cohorts and 15 healthy control subjects with normal hepatic function (Cohort D). Enrollment of 8 subjects with mild hepatic impairment (Cohort A) proceeded only if there is evidence of reduced clearance of aramchol in Cohort B. Assignment to cohorts A to C, was according to Child Pugh classification system.

Serial blood samples for PK analysis of aramchol concentrations in plasma were collected before dosing (0 hour) and up to 168 hours for healthy subjects and 240 hours for hepatically impaired subjects after administration of aramchol.

In Part 2 (multiple-dose), a cohort of 4 subjects comprising of mild, 7 moderate , as well as a cohort of 7 healthy volunteers was administered with aramchol as multiple doses to obtain the PK profile of aramchol at steady state. Aramchol was given twice daily for 12 days. Trough blood samples for analysis of aramchol plasma concentrations was collected before the AM dose on several days and at intervals to 12 hours after the AM dose on Day 12.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female 18 to 79 years of age, inclusive.
2. The subject has a body mass index of 19 to 40 kg/m2, inclusive, at screening.
3. Females of childbearing potential must practice a highly effective method of contraception throughout the study period and for 1 month after treatment discontinuation.
4. Male subjects with female partners of childbearing potential must be vasectomized, be willing to use an acceptable method of birth control, or practice abstinence during the study.
5. The subject has a resting pulse rate of ≥40 and <100 beats per minute with no clinically significant deviation as judged by the investigator.
6. The subject has a QT interval corrected for heart rate using Fridericia's formula of <500 msec.
7. The subject agrees to comply with all protocol requirements.
8. The subject is able to provide written informed consent.

   Additional Inclusion Criteria for Healthy Subjects Only (Cohort D):
9. The subject has normal hepatic function.
10. The subject has a resting blood pressure of 90 to 150 mm Hg (systolic) and 50 to 100 mm Hg (diastolic).
11. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings.

    Additional Inclusion Criteria for Subjects With Hepatic Impairment Only (Cohorts A, B, and C):
12. The subject has cirrhosis with evidence of impaired liver function. The etiology of the cirrhosis may be alcoholic, autoimmune, nonalcoholic steatohepatitis, or chronic viral hepatitis type B or C.
13. The subject has chronic (more than 6 months) and stable hepatic impairment (ie, no acute episodes of illness within 30 days before screening due to deterioration of hepatic function) as assessed by a Child-Pugh classification score of mild (5 to 6 points), moderate (7 to 9 points), or severe (10 to 15 points).
14. The subject has a resting blood pressure of 90 to 155 mm Hg (systolic) and 50 to 100 mm Hg (diastolic).
15. The subject is judged by the investigator to be in good general health, as determined by medical history, clinical laboratory assessments, vital sign measurements, 12 lead ECG results, and physical examination findings, except for findings that, as judged by the investigator, are consistent with the subject's hepatic impairment or other stable concomitant medical conditions.

Exclusion Criteria:

1. The subject has a history or clinical manifestations of a significant neurological, renal, cardiovascular, gastrointestinal, pulmonary, hematologic, immunologic, or psychiatric disease that would preclude study participation, as judged by the investigator.
2. The subject has a positive test result for human immunodeficiency virus type 1 or 2 antibodies at screening.
3. The subject has a history of drug abuse within 3 months before screening.
4. The subject has a history of alcoholism within 3 months before screening, or excessive alcohol consumption (regular alcohol intake >15 units per week) (1 unit is equal to approximately ½ pint [200 mL] of beer, 1 small glass [100 mL] of wine, or 1 measure [25 mL] of spirits).
5. The subject smokes >10 cigarettes daily and is unwilling to reduce to <5 daily from the time of screening through the last PK sample.
6. The subject is unable or unwilling to abstain from alcohol, caffeine, xanthine containing beverages or food (eg, coffee, tea, chocolate, and caffeinated sodas, colas), grapefruit, grapefruit juice, Seville oranges, or products containing any of these, from 48 hours prior to study drug dosing until discharge.
7. The subject is involved in strenuous activity or contact sports within 24 hours of the first dose of study drug or during the study.
8. The subject has donated blood or blood products >450 mL within 3 months before the first dose of study drug.
9. The subject has a presence or history of relevant drug and/or food allergies (ie, allergy to aramchol, cholic acid, or any excipients, or any significant food allergy.
10. The subject has received study drug in another investigational study within 30 days of dosing.
11. In the opinion of the investigator, the subject is not suitable for entry into the study.

For additional exclusion criteria specific to hepatic impaired subjects and healthy volunteers, see protocol.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Gilgun-Sherki, PhD, MBA, Study Director — Executive Drug Development Consultant
Locations (3):
- United States (3):
  - Division of Clinical Pharmacology, University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Alliance for Multispecialty Research, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Mild Hepatic Impairment (Cohort A): 8 mild hepatic impaired subjects
  Aramchol 600mg single dose: aramchol acid tablet 600mg, single dose
- Part 1: Moderate Hepatic Impairment (Cohort B): 8 moderate hepatic impaired subjects
  Aramchol 600mg single dose: aramchol acid tablet 600mg, single dose
- Part 1: Severe Hepatic Impairment (Cohort C): 8 severe hepatic impaired subjects
  Aramchol 600mg single dose: aramchol acid tablet 600mg, single dose
- Part 1: Healthy Volunteers (Cohort D): 15 matched healthy volunteers
  Aramchol 600mg single dose: aramchol acid tablet 600mg, single dose
- Part 2: Mild Hepatic Impairment Cohort: 4 hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
- Part 2- Moderate Hepatic Impairment Cohort: 7 hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
- Part 2: Healthy Volunteers Cohort: 7 matched healthy volunteers
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
Period: Overall Study
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2- Moderate Hepatic Impairment Cohort | Part 2: Healthy Volunteers Cohort
Started | 8 | 8 | 8 | 15 | 4 | 7 | 7
Completed | 8 | 8 | 8 | 15 | 4 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population in Part 1 included mild hepatic impairment subjects, moderate hepatic impairment subjects, severe hepatic subjects, and healthy matched control subjects. Population in Part 2 included mild hepatic impairment subjects, moderate hepatic impairment subjects, and healthy matched control subjects.
Groups:
- Part 2: Mild Hepatic Impairment Cohort: 4 mild hepatic impaired subjects (mild, moderate or severe)
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
- Part 2: Moderate Hepatic Impairment Cohort: 7 moderate hepatic impaired subjects (mild, moderate or severe)
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
- Total: Total of all reporting groups
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Hepatic Impairment Cohort | Part 2: Healthy Volunteers Cohort | Total
Number analyzed (Participants) | 8 | 8 | 8 | 15 | 4 | 7 | 7 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 5 | 10 | 2 | 4 | 6 | 39
  >=65 years | 1 | 3 | 3 | 5 | 2 | 3 | 1 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (8.10) | 63.3 (9.02) | 62.0 (6.35) | 59.7 (8.50) | 64.0 (4.16) | 60.1 (8.47) | 60.1 (6.82) | 60.86 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 4 | 1 | 1 | 2 | 16
  Male | 7 | 5 | 4 | 11 | 3 | 6 | 5 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 1 | 1 | 1 | 3 | 3 | 13
  Not Hispanic or Latino | 8 | 4 | 7 | 14 | 3 | 4 | 4 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 7
  White | 5 | 8 | 8 | 10 | 2 | 7 | 6 | 46
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 15 | 4 | 7 | 7 | 57
Child-Pugh total scores [Mean (Standard Deviation); unit: points] — The Child-Pugh score uses 5 clinical measures (i.e., total bilirubin, serum albumin, prothrombin time, ascites, and hepatic encephalopathy) to assess liver disease. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe (score<5- not liver disease)
  Class A
  * 5 to 6 points
  * least severe liver disease
  * one- to five-year survival rate: 95 percent
  Class B
  * 7 to 9 points
  * moderately severe liver disease
  * one- to five-year survival rate: 75 percent
  Class C
  * 10 to 15 points
  * most severe liver disease
  * one- to five-year survival rate: 50 percent Population: Healthy volunteers don't have any meaningful disease, and thus they don't have any liver disease or liver issues and as a result they don't have a Child-Pugh score
  points
    number analyzed (Participants) | 8 | 8 | 8 | 0 | 4 | 7 | 0 | 35
    (all) | 5.38 (0.518) | 8.25 (0.886) | 11.50 (1.512) |  | 5.75 (0.5) | 7.71 (0.756) |  | 7.94 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tau, Steady State
Description: AUC from time 0 to the dosing interval tau measured at steady state.
  Blood was collected at the following time points: before dosing (0 hour) and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 48, 72, 96, 120, 144, 168, 192, and 240 hours
Time Frame: Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h•ng/mL
Groups:
- Part 2: Moderate Impairment Cohort: 7 hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Impairment Cohort | Part 2: Healthy Volunteers Cohort
Number analyzed (Participants) | 8 | 8 | 8 | 15 | 4 | 7 | 7
h•ng/mL | 96100 (138.29) | 107000 (154.13) | 103000 (148.09) | 69500 (0) | 63300 (4.3) | 55900 (31.4) | 61400 (26)

2. Primary Outcome: Cmax,ss
Description: Maximum plasma concentrations (Cmax,ss)
  Blood was collected at the following time points: before dosing (0 hour) and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 48, 72, 96, 120, 144, 168, 192, and 240 hours
Time Frame: Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Hepatic Impairment Cohort | Part 2: Healthy Volunteers Cohort
Number analyzed (Participants) | 8 | 8 | 8 | 15 | 4 | 7 | 7
ng/mL | 1950 (138.17) | 1890 (134.26) | 1480 (105.22) | 1410 (0) | 5750 (5.2) | 5380 (26.1) | 6040 (21.3)

3. Primary Outcome: Apparent Total Oral Clearance, Single Dose
Description: CL/F measured after single dose in Part 1
  Blood was collected at the following time points: before dosing (0 hour) and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 48, 72, 96, 120, 144, 168, 192, and 240 hours
Time Frame: Day 11
Population: Note that apparent total oral clearance data was analyzed for Part 1 only, where comparison was made between Healthy volunteers and Hepatic impairment patients. Such data was not collected and analyzed for Part 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Part 2: Mild Hepatic Impairment Cohort: 4 mild hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
- Part 2: Moderate Impairment Cohort: 7 moderate hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Impairment Cohort | Part 2: Healthy Volunteers Cohort
Number analyzed (Participants) | 8 | 8 | 8 | 15 | 0 | 0 | 0
L/h | 5.96 (43.8) | 5.23 (29.2) | 5.86 (52.5) | 8.01 (50.1) |  |  |

4. Secondary Outcome: Number of Subjects With Significant TEAEs
Description: The number of significant treatment-related adverse events
Time Frame: Part 1: up to 22 days; Part 2: up to 27 days
Population: All subjects
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Moderate Hepatic Impairment Cohort: 7 mild hepatic impaired subjects
  Aramchol 300mg, bid: aramchol acid tablet 300mg, bid for 12 days
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Hepatic Impairment Cohort | Part 2: Healthy Volunteers Cohort
Number analyzed (Participants) | 8 | 8 | 8 | 15 | 4 | 7 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time the subject signed the informed consent until study completion (i.e., End of study- 30 days).
Arm/Group | Part 1: Mild Hepatic Impairment (Cohort A) | Part 1: Moderate Hepatic Impairment (Cohort B) | Part 1: Severe Hepatic Impairment (Cohort C) | Part 1: Healthy Volunteers (Cohort D) | Part 2: Mild Hepatic Impairment Cohort | Part 2: Moderate Impairment Cohort | Part 2: Healthy Volunteers Cohort
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/15 | 0/4 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/15 | 0/4 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/15 | 0/4 | 1/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Mild Hepatic Impairment (Cohort A) (N=8) | Part 1: Moderate Hepatic Impairment (Cohort B) (N=8) | Part 1: Severe Hepatic Impairment (Cohort C) (N=8) | Part 1: Healthy Volunteers (Cohort D) (N=15) | Part 2: Mild Hepatic Impairment Cohort (N=4) | Part 2: Moderate Impairment Cohort (N=7) | Part 2: Healthy Volunteers Cohort (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT04480827/Prot_SAP_000.pdf